CLINICAL TRIAL: NCT03110003
Title: Comparing Low-dose Bupivacaine With Epidural Volume Extension to Standard Bupivacaine Dosing for Short Obstetric Procedures: A Prospective, Randomized Study
Brief Title: Bupivacaine With Epidural Volume Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Mark Powell, Assistant Professor, University of Alabama at Birmingham
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: F1605020005
Record Dates: First submitted 2017-03-30; First posted 2017-04-12 (Actual); Results first posted 2018-09-13 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-11

CONDITIONS: Spinal Anesthesia; Epidural; Anesthesia
Keywords: Neuraxial epidural techniques; Combined spinal epidural; Epidural volume extension; Transient Neurologic Symptoms (TNS)
MeSH Terms: interventions — Bupivacaine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- 10 mg Bupivacaine (Active Comparator): Subjects will receive 10 mg of preservative-free isobaric bupivacaine with 12.5mcg of fentanyl.
  Interventions: Drug: 10 mg Bupivacaine
- 5 mg Bupivacaine (Active Comparator): Subjects will receive 5 mg of preservative-free isobaric bupivacaine with 12.5mcg of fentanyl in combination with 10 mL of sterile saline injected into the epidural space.
  Interventions: Drug: 5 mg Bupivacaine

INTERVENTIONS:
Drug: 10 mg Bupivacaine — 10 mg of preservative-free isobaric bupivacaine with 12.5mcg of fentanyl injected to the epidural space
  Other Names: Marcaine and Sensorcaine
  Arms: 10 mg Bupivacaine
Drug: 5 mg Bupivacaine — 5 mg of preservative-free isobaric bupivacaine with 12.5mcg of fentanyl in combination with 10 mL of sterile saline injected into the epidural space.
  Other Names: Marcaine and Sensorcaine
  Arms: 5 mg Bupivacaine

SUMMARY:
In this study the investigator will address the efficacy of using low dose bupivacaine spinal anesthesia (SA) in combination with epidural volume extension (EVE) for patients undergoing short obstetric procedures.

DETAILED DESCRIPTION:
Due to risks to both the mother and fetus, neuraxial anesthesia - spinal, epidural, or combined spinal-epidural (CSE) - is preferred over general anesthesia for all obstetrical procedures. However, one downside to neuraxial anesthesia is the increased time patients have to stay in the post-anesthesia care unit (PACU) due to residual numbness from the neuraxial block. In this study, the investigators will address the efficacy of using low dose bupivacaine spinal anesthesia (SA) in combination with epidural volume extension (EVE) for patients undergoing short obstetric procedures. This will be accomplished by performing a CSE with: 1) injecting the local anesthesia in the spinal space; 2) injecting sterile saline into the epidural space to help increase the spread of the local anesthesia in the spinal space. The idea is that physicians will be able to use less local anesthetic due to getting a greater spread of medication. This lower amount of local anesthetic will lead to a decreased duration of the spinal block; therefore, it will significantly decrease PACU length of stay. This technique will be compared to our traditional dose of spinal anesthetic without EVE in the CSE. Both groups will have an epidural catheter in place to allow us to give any additional local anesthetic to keep the patient comfortable throughout the procedure if the spinal anesthesia begins to wear off. The aim of this study is to determine if low dose spinal bupivacaine in conjunction with EVE can decrease the PACU recovery time for short obstetric procedures while still providing an adequate surgical block.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing short obstetric procedure in the operating room requiring neuraxial anesthesia.

Exclusion Criteria:

* coagulopathy
* platelets <80,000
* allergy to local anesthetic or fentanyl
* previous spinal surgery
* spinal or intracranial mass
* history of lower extremity weakness

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 45 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-12-01 (Actual); Study Completion 2018-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Powell, MD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- UAB Department of Anesthesiology and Perioperative Medicine, Birmingham, Alabama, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Started | 21 | 24
Completed | 21 | 24
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine | Total
Number analyzed (Participants) | 21 | 24 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 21 | 24 | 45
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 21 | 24 | 45
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 21 | 24 | 45

OUTCOME MEASURES:

1. Primary Outcome: Time Until PACU Discharge in Minutes
Description: Time from entrance into the PACU until PACU discharge criteria met
Time Frame: Baseline up to 48 hrs postoperatively
Measure: Median (Full Range); unit: minutes
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Number analyzed (Participants) | 21 | 24
minutes | 135 [103 to 182.5] | 50 [42 to 57.5]

2. Secondary Outcome: Peak Block Height
Description: Thoracic dermatome level as assessed by pinprick
Time Frame: Baseline up to 3 hours
Population: Thoracic dermatome level as assessed by pinprick
Measure: Median (Inter-Quartile Range); unit: Thoracic dermatome
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Number analyzed (Participants) | 21 | 24
Thoracic dermatome | 5 [4 to 7.5] | 5 [3.25 to 7.75]

3. Secondary Outcome: Degree of Peak Motor Blockade by Modified Bromage Scale
Description: Motor blockade will be determined by the patient's ability to lift her legs
  This is simple scale used to assess motor function in the patients' legs. A numerical value from 0 to 4 is assigned to visual inspection of how well the patient can move her legs. 0=ability to maintain a leg lift for prolonged periods; 1=ability to lift legs briefly; 2=ability to bend knees; 3=ability to wiggle toes; 4=no movement in legs. A score of 0 means complete movement (no blockade) in the legs, whereas a score of 4 means no movement (complete blockade) in the legs.
Time Frame: Baseline up to 3 hours
Measure: Mean (Inter-Quartile Range); unit: score on a scale
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Number analyzed (Participants) | 21 | 24
score on a scale | 3 [3 to 4] | 3 [2 to 3]

4. Secondary Outcome: Time Elapsed Until Motor Block Regresses to Modified Bromage Score = 0
Description: Time until score of <2 reached on Modified Bromage scale
  This is simple scale used to assess motor function in the patients' legs. A numerical value from 0 to 4 is assigned to visual inspection of how well the patient can move her legs. 0=ability to maintain a leg lift for prolonged periods; 1=ability to lift legs briefly; 2=ability to bend knees; 3=ability to wiggle toes; 4=no movement in legs. A score of 0 means complete movement (no blockade) in the legs, whereas a score of 4 means no movement (complete blockade) in the legs. Once the patient received as score of 0, the time ended. Again, 0=ability to maintain a leg lift for prolonged periods.
Time Frame: Baseline up to 6 hours
Population: Time elapsed until motor block regresses to modified Bromage = 0.
Measure: Median (Inter-Quartile Range); unit: Minutes
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Number analyzed (Participants) | 21 | 24
Minutes | 181 [141 to 225.5] | 66 [44.5 to 87]

5. Secondary Outcome: Quality of Block as Determined by Subjective Pain Assessment
Description: Determined by any pain reported during surgery and/or the need to supplement through the epidural
Time Frame: Baseline up to 6 hours
Population: Quality of Block as determined by subjective pain assessment was not collected by the investigators.
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Number analyzed (Participants) | 0 | 0

6. Secondary Outcome: Patient Satisfaction as Determined by a Likert-type Scale
Description: Patient satisfaction of a scale of 1-10
  This scale is grade from 1 to 10 with 1 being "highly dissatisfied" with the anesthetic technique and 10 being "highly satisfied." Each patient was asked to rate their experience with the anesthetic technique provide. They could choose any number between 1 and 10. Numbers close to 10 represented a higher satisfaction with the anesthetic technique.
Time Frame: At 6 hrs postoperatively
Population: Patient satisfaction as determined by a Likert-type scale was not collected by the investigators.
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 2 years
Arm/Group | 10 mg Bupivacaine | 5 mg Bupivacaine
All-Cause Mortality (participants affected / at risk) | 0/21 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/21 | 0/24
Other Adverse Events (participants affected / at risk) | 0/21 | 0/24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03110003/Prot_SAP_000.pdf